CLINICAL TRIAL: NCT00310336
Title: Chronic Hepatitis C: Treatment of (Peg)Interferon Alpha - Ribavirin Non-Responders With Pegylated Interferon alpha2b, Ribavirin, AdoMet and Betaine
Brief Title: Chronic Hepatitis C Non-Responder Study With AdoMet and Betaine
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EKBB 37/06
Record Dates: First submitted 2006-03-31; First posted 2006-04-03 (Estimated); Last update posted 2010-10-28 (Estimated); Status verified 2010-10

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — S-Adenosylmethionine; Betaine; peginterferon alfa-2b; Ribavirin

INTERVENTIONS:
Drug: S-adenosyl-L-methionine
Drug: betaine
Drug: pegylated interferon alpha2b
Drug: ribavirin

SUMMARY:
50-60% of patients with chronic hepatitis C are not cured by treatment with pegylated IFNα plus ribavirin.

Retreatment of non-responders of previous (pegylated) IFNα plus ribavirin therapies with pegylated IFNα plus ribavirin results in a sustained response in less than 10% of the patients.

Extensive analysis of IFNα signaling in cells expressing HCV proteins, in transgenic mice expressing HCV proteins, and in liver biopsies from patients with chronic hepatitis C point to STAT1 methylation as an important posttranslational modification targeted by HCV to inhibit IFNα signaling.

STAT1 methylation can be increased and IFNα can be improved by adding AdoMet and betaine.

The study is designed to test the hypothesis that a combination treatment with pegylated IFNα2b, ribavirin, AdoMet and betaine is superior to the current standard combination therapy with pegylated IFNα plus ribavirin.

ELIGIBILITY:
Inclusion Criteria:

* Male and female between 18 and 65 years.
* Non-responders in previous treatments with IFNα plus ribavirin or pegylated IFNα plus ribavirin.
* Elevated ALT-levels on at least two occasions during >6 months preceding entry.
* Detection of HCV RNA in serum (PCR).
* Compensated liver disease (Child-Pugh A) and a Child-Pugh score <5.
* The following minimal hematologic and biochemical criteria:
* Hemoglobin for males and females >11g/dl
* Absolute Neutrophil count >1500 cells/mm3
* Platelets >75'000/mm3
* HBs Ag negative.
* ANA <1:320, and no evidence for autoimmune hepatitis.
* α-Fetoprotein <50μg/l (when between upper limit of normal and 50μg/l, ultrasonographical exclusion of hepatocellular carcinoma (HCC) is needed).
* Fasting blood glucose within normal limits, if history of diabetes or hypertension, a pre-therapy ocular examination is indicated.
* TSH within normal limits or adequately controlled.
* Negative urine or blood pregnancy test (for women of childbearing potential) documented within the 2-3 week period prior to the first dose of study drug. Additionally, all fertile males and females must be using effective contraception during treatment and during the 6 months after treatment end. This may include, but is not limited to, using birth control pills, IUDs, condoms, diaphragms, or implants, being surgically sterilized, or being in a post-menopausal state.
* Willingness to give written informed consent and willingness to participate to and comply with the study

Exclusion Criteria:

* Women with ongoing pregnancy or breast feeding.
* Positive test at screening for anti-HAV IgM Ab, HBsAg, anti-HBc IgM Ab, HBe Ag.
* Positive test at screening for HIV.
* History or other evidence of a medical condition associated with chronic liver disease other than HCV (e.g., hemochromatosis, autoimmune hepatitis, alcoholic liver disease, toxin exposures).
* Hypersensitivity to study drugs.
* Participation in any other clinical trial within 30 days of entry into this protocol.
* Treatment with any investigational drug within 30 days of entry into this protocol.
* History or evidence of decompensated liver disease (Child-Pugh B/C) and a Child-Pugh score >5. Ascites, coagulopathy, hyperbilirubinemia, hepatic encephalopathy, or hypoalbuminemia and a Child-Pugh score >5 are conditions consistent with decompensated liver disease.
* History or other evidence of bleeding from esophageal varices or other conditions consistent with decompensated liver disease.
* Hepatocellular carcinoma (HCC) or α-Fetoprotein >50μg/l.
* Patients with organ transplants other than cornea and hair transplant.
* Therapy with any antisystemic or immunomodulatory treatment (including supra-physiologic doses of steroids or radiation) <6 months prior the first dose of study drug
* Hemoglobinopathy (e.g. thalassemia) or any other cause of or tendency for hemolysis.
* Any known preexisting medical condition that could interfere with the patient's participation in and completion of the study such as:
* Preexisting psychiatric condition, especially depression, or a history of severe psychiatric disorder, such as major psychosis, suicidal ideation and/or suicidal attempts (based on a mandatory psychiatric advice).
* CNS trauma or active seizure disorders requiring medication.
* Significant cardiovascular dysfunction.
* Poorly controlled diabetes mellitus.
* Renal dysfunction, i.e. serum creatinine levels >1.5 times upper limit of normal.
* Autoimmune diseases.
* Evidence of severe retinopathy (e.g. CMV retinitis, macular degeneration).
* Any medical condition requiring, or likely to require during the course of the study, chronic systemic administration of steroids.
* Clinical gout.
* Important substance abuse (alcohol >80 g/d, i.v. drugs etc.).
* Active opportunistic infections.
* Non-Hodgkin lymphoma or Hodgkin lymphoma.
* Kaposi sarcoma.
* Inability or unwillingness to provide informed consent or abide by the requirements of the study.
* Male partners of pregnant women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2006-08; Primary Completion 2009-08 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Sustained response rate

SECONDARY OUTCOMES:
Early virologic response after 12 weeks of therapy with PegIntron, Rebetol, AdoMet and betaine.

CONTACTS AND LOCATIONS:
Overall Officials: Markus H Heim, MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Canton of Basel-City, Switzerland

REFERENCES:
- [Background] Duong FH, Christen V, Filipowicz M, Heim MH. S-Adenosylmethionine and betaine correct hepatitis C virus induced inhibition of interferon signaling in vitro. Hepatology. 2006 Apr;43(4):796-806. doi: 10.1002/hep.21116. PMID 16557551
- [Background] Duong FH, Christen V, Berke JM, Penna SH, Moradpour D, Heim MH. Upregulation of protein phosphatase 2Ac by hepatitis C virus modulates NS3 helicase activity through inhibition of protein arginine methyltransferase 1. J Virol. 2005 Dec;79(24):15342-50. doi: 10.1128/JVI.79.24.15342-15350.2005. PMID 16306605
- [Background] Duong FH, Filipowicz M, Tripodi M, La Monica N, Heim MH. Hepatitis C virus inhibits interferon signaling through up-regulation of protein phosphatase 2A. Gastroenterology. 2004 Jan;126(1):263-77. doi: 10.1053/j.gastro.2003.10.076. PMID 14699505
- [Background] Blindenbacher A, Duong FH, Hunziker L, Stutvoet ST, Wang X, Terracciano L, Moradpour D, Blum HE, Alonzi T, Tripodi M, La Monica N, Heim MH. Expression of hepatitis c virus proteins inhibits interferon alpha signaling in the liver of transgenic mice. Gastroenterology. 2003 May;124(5):1465-75. doi: 10.1016/s0016-5085(03)00290-7. PMID 12730885
- [Background] Heim MH, Moradpour D, Blum HE. Expression of hepatitis C virus proteins inhibits signal transduction through the Jak-STAT pathway. J Virol. 1999 Oct;73(10):8469-75. doi: 10.1128/JVI.73.10.8469-8475.1999. PMID 10482599
- [Derived] Filipowicz M, Bernsmeier C, Terracciano L, Duong FH, Heim MH. S-adenosyl-methionine and betaine improve early virological response in chronic hepatitis C patients with previous nonresponse. PLoS One. 2010 Nov 8;5(11):e15492. doi: 10.1371/journal.pone.0015492. PMID 21079746